CLINICAL TRIAL: NCT04555083
Title: Relationship Between Chronic Ankle Instability and Sacroiliac Joint Dysfunction
Brief Title: Association Between Chronic Ankle Instability and Sacroiliac Joint Dysfunction
Status: Completed | Type: Observational
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Dalia Mohammad Mohammad Mosaad, Principal investigator, Cairo University
Other Study IDs: P.T.REC/012/002302
Record Dates: First submitted 2020-09-14; First posted 2020-09-18 (Actual); Last update posted 2021-06-08 (Actual); Status verified 2021-06

CONDITIONS: Sacroiliac Joint Dysfunction
Keywords: chronic ankle instability; Sacroiliac joint dysfunction

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- CAI group: Case group is CAI group that recruit patients complain of ankle insatiability and giving way mainly
- control group: control group recruits participants with non injured ankle, matched with case group in gender and dominant limb

SUMMARY:
chronic ankle instability previously approved in many studies that it may lead to more proximal adaptations and negative long term consequences. one of those studies reported, ankle instability patients has hamstring muscle shortening in comparison with non sprained subjects. another one concluded that gluteus maximums muscle has delayed activation and weakness in CAI patients. Both muscles (hamstring and gluteus Maximus ) contribute to sacroiliac joint stability. therefore, this study asked a novel research question, was sacroiliac joint dysfunction (SIJD) associated with CAI?

DETAILED DESCRIPTION:
The sample size of this study had been calculated based on the primary outcome that was the association between CAI and SIJD after a pilot study done in order to detect odd's ratio. , calculation made by a program developed by the Centers for Disease Control and Prevention with the following inputting data :

Two-sided confidence interval 95%, power 80%, ratio of controls to cases 1, percent of control exposed 4.5% , odds ratio 32%. The sample size calculations required for this study was 28 participants (14 in each group).

Data distributions was checked for normality using Shapiro-Wilk test and for equality of variance using Box's test. Box and whiskers plots were used for detecting the outliers. Descriptive statistics calculated for demographic data. Intraclass correlation coefficients (ICC) and standard errors of measurement (SEM) were calculated to estimate the intratester reliability and precision of measurement for the static pelvic rotation

The outcomes of these study were:

1. Association between CAI and SIJD represents through odd's ratio (primary outcome)
2. Pelvic torsion difference between CAI and control Calculated by Mann- Whitney test (secondary outcome)
3. Correlations between pelvic torsion with perceived ankle instability and number of giving way episodes calculated Pearson correlation coefficient(secondary outcome) Effect size analysis was calculated to determine the clinical significant difference. Statistical analysis was conducted using the statistical package for social studies (SPSS) for windows, version 24 (SPSS, Inc., Chicago, IL). The normative data presented as Mean ± standard deviation (SD) while non-normative data presented as median. Significance was set at p < 0.05 and total study power was set 80%

ELIGIBILITY:
Inclusion Criteria:

1. young active people between 18-30 years old
2. CAI group has a self-report of a past history of unilateral ankle inversion injury since at least more than 1 year before the study onset
3. Required a period of protected weight bearing and/or immobilization at least one day
4. The patient reported a tendency to give way or repeatedly turn over during functional activity
5. At least 2 giving way episodes during the year before the study onset and/or recurrent ankle sprain
6. Perceived that the ankle was chronically weaker, more painful, and/or less functional than other non-injured ankle or than before first injury.
7. Positive anterior drawer test and /or talar tilt test

Exclusion Criteria:

* Exclusion Criteria for both groups (CAI and Control )

  1. Trunk asymmetry angle 5 - 7 degrees
  2. Leg length difference more than 0.5 cm
  3. History of autoimmune diseases, complains of ankylosing spondylitis and morning stiffness
  4. Participation in physical therapy regimen within a year before enrolling in the study
  5. Bilateral ankle sprain injury
  6. Ankle sprain within 3 months of participation
  7. If they had only midline or symmetrical pain above the level of L5 or radicular pain with neurological deﬁcits (sensory or motor deﬁcits)
  8. History of spinal surgery, infection, tumors, fracture of the spine, pelvis or lower extremities within 2 years before enrolling in the study.
  9. Hospitalization for severe trauma or car accident
  10. Pregnant women
  11. Any neurological and orthopedics diseases could affect the conditions

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Recruited from faculty of physical therapy through announcements for volunteering to participate in noninvasive study include patients complaining of ankle instability and others did not have any injury in their ankle before
Sampling Method: Non-Probability Sample
Enrollment: 45 (Actual)
Dates: Start 2020-01-03 (Actual); Primary Completion 2020-09-30 (Actual); Study Completion 2020-11-30 (Actual)

PRIMARY OUTCOMES:
odd's ratio of sacroiliac joint dysfunction | throughout the study about 1 year
  association between CAI and sacroiliac joint dysfunction

SECONDARY OUTCOMES:
difference of pelvic torsion between CAI and control | throughout the study about 1 year
  pelvic torsion is pelvic asymmetry in sagittal plane
correlation between pelvic torsion and giving way episodes | throughout the study about one year
  giving way episodes throughout the previous year and pelvic torsion by inclinometer
corelation between pelvic torsion and perceived sensation of instability | throughout the study about 1 year
  pelvic torsion by inclinometer and perceived instability sensation through visual analogue scale, ranged from 0-10 with high score means worse result

CONTACTS AND LOCATIONS:
Overall Officials: Dalia mossad, professor, Principal Investigator — professor at faculty of physical therapy Cairo university
Locations (1):
- ‪Afaf Tahoon‬, Dokki, Giza Governorate, Egypt